CLINICAL TRIAL: NCT02746913
Title: Ambulatory Pessary Trial as a Preoperative Method for Diagnosing Occult Stress Urinary Incontinence
Brief Title: Ambulatory Pessary Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-00598
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Urinary Incontinence
Keywords: Pelvic, Urodynamic, Vaginal Wall
MeSH Terms: conditions — Urinary Incontinence | interventions — Pessaries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Urodynamics, followed by Pessary (Experimental)
  Interventions: Device: Urodynamics; Device: Pessary
- Pessary, followed by Urodynamics (Experimental)
  Interventions: Device: Urodynamics; Device: Pessary

INTERVENTIONS:
Device: Urodynamics — Urodynamics is performed with the Aquarius XT Laborie system and a fluoroscopic images are obtained with a GE OCE 9800 c-arm fluoroscopy unit. Urodynamic testing will be performed in a seated position with a pessary from the ambulatory pessary trial in place. Post residual void will be measured at the start of the urodynamics.
Device: Pessary — A pessary is a silicone disc that is used in to support the uterus and vagina of women with vaginal prolapse. During this study, the pessary that will be used is a ring with support. This is a disc shape with a membrane stretched across the center. It is a device used in standard practice and is safe to keep in place for up to 3 months at a time. The subjects will be fit with a pessary asked to wear the pessary for 3 days.

SUMMARY:
The purpose of this study is to compare two methods for assessing patients with pelvic organ prolapse for occult stress urinary incontinence. Urodynamic testing is the most widely accepted and well-studied method for diagnosing occult stress urinary incontinence preoperatively, but an ambulatory pessary trial is a less expensive option that is available to a wider group of practitioners and evaluates patient while they are engaged in their daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Patients planning to undergo pelvic organ prolapse surgery and preoperative urodynamic testing within 6 months of recruitment.
* Stage 2 or greater pelvic organ prolapse on pre op POP-Q exam
* Negative stress test on clinical exam
* Cognitive capacity to complete questionnaires and voiding diary

Exclusion Criteria:

* Stress incontinence during provocative stress test on pre-operative exam.
* Occult stress urinary incontinence demonstrated on pre-operative physical exam
* Known ability to retain a pessary for the 3 day trial
* < age 18
* History of bladder augmentation or artificial sphincter
* Known neurologic disease effecting bladder (spinal cord injury, Multiple Sclerosis, Parkinson's Disease, etc.)
* Non ambulatory patients
* Active infections of the vagina or pelvis (Pelvic inflammatory disease, infectious vaginitis, etc.)
* Occult stress urinary incontinence demonstrated on pre-operative physical exam
* Known ability to retain a pessary for the 3 day trial
* < age 18
* History of bladder augmentation or artificial sphincter
* Known neurologic disease effecting bladder (spinal cord injury, Multiple Sclerosis, Parkinson's Disease, etc.)
* Non ambulatory patients
* Active infr

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Medical, Epidemiological, and social Aspects of Aging (MESA) questionnaire | 3 Days
  leakage on a voiding diary.
Overactive bladder quality of life (QAB-Q)- short term questionnaire | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Brucker, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States